CLINICAL TRIAL: NCT00049335
Title: Protocol For Assessment Of Capecitabine For Advanced Colorectal Cancer In Patients Aged 70 Years And Older (And In A Cohort Of Patients Younger Than 60 Years)
Brief Title: S0030: Capecitabine in Treating Older Patients W/Metastatic or Recurrent Colorectal Cancer That Cannot Be Surgically Removed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258049; S0030 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine (Experimental): Capecitabine 1,000 mg/m^2/dose (2,000 mg/m^2/day) BID, PO, Days 1-14 of 21 day cycle.
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: capecitabine — 1,000 mg/m^2/dose (2,000 mg/m^2/day) BID, PO, on Days 1-14 of 21 day cycle
  Other Names: NSC-712807

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of capecitabine in treating older patients who have metastatic or recurrent colorectal cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of enrolling patients aged 70 and over with unresectable metastatic or recurrent colorectal cancer to a structured phase II study.
* Determine the anticancer efficacy of capecitabine, in terms of objective response rate (confirmed and unconfirmed, complete and partial responses) and 2-year survival, in these patients.
* Determine the toxicity and tolerability of this drug in these patients.
* Determine the feasibility of using standardized self-report measures of comorbidity, depression, and functional status of patients treated with this drug.
* Determine the clinical pharmacology of this drug in these patients.
* Determine whether patients under 60 years of age treated with this drug have clinical pharmacologic parameters similar to those reported in the literature.

OUTLINE: This is a multicenter study. Patients are stratified according to age (70 and over vs 18 to 59).

Patients receive oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 80 patients (60 patients aged 70 and over, 20 patients aged 18 to 59) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or recurrent colorectal cancer not amenable to surgical resection
* Measurable disease
* No known brain metastases by MRI or CT scan

PATIENT CHARACTERISTICS:

Age

* 70 and over OR
* 18 to 59

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT (serum glutamate oxaloacetate transaminase) or SGPT (serum glutamate pyruvate transaminase) no greater than 2 times ULN

Renal

* Creatinine no greater than 2 times ULN
* Creatinine clearance greater than 50 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No known seizure disorder
* No other malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, adequately treated stage I or II cancer currently in complete remission, or any other cancer for which the patient has been disease free for 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for advanced cancer
* Prior adjuvant chemotherapy allowed provided recurrence occurred more than 1 year after the last treatment

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 4 weeks since prior sorivudine or brivudine
* No concurrent sorivudine or brivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrolling patients aged 70 years or older to a Phase II trial including pharmacokinetic sampling | Registration

SECONDARY OUTCOMES:
Efficacy of capecitabine for management of advanced colorectal cancer patients aged 70 years or older based on objective response rate and 2 year survival | 2 years
Toxicity | 3 years
Assess parameters of clinical pharmacology of capecitabine in patients aged 70 years or older including half life value(s), AUC (area under curve) and steady state levels | 3 years
Assess whether patients under 60 years have clinical pharmacologic parameters similar to those reported in the literature | 3 years
Explore, at a preliminary level, the feasibility of studying genetic polymorphisms and gene expression levels of enzymes involved in drug metabolism and resistance to capecitabine | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Study Chair — University of Southern California
Locations (90):
- United States (90):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington